CLINICAL TRIAL: NCT07264465
Title: A Clinical Trial to Evaluate the Effects of a Chickpea Pasta on Gut Health, Blood Glucose, and Overall Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Banza LLC (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20724
Record Dates: First submitted 2025-09-30; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Gut Health; Gastrointestinal Health
Keywords: Microbiome Diversity; Nutritional Supplement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chickpea Pasta Intervention Arm (Experimental): Participants will consume 1½ cups (188g) of cooked Banza chickpea pasta once daily, 5 days per week, for 12 weeks.
  Interventions: Dietary Supplement: Chickpea Pasta

INTERVENTIONS:
Dietary Supplement: Chickpea Pasta — The intervention is intended to assess the effects of a high-fiber, legume-based dietary product on gut microbiome diversity, gastrointestinal function, and metabolic biomarkers.

SUMMARY:
This is a single-arm, 12-week pilot study evaluating the effects of a chickpea pasta on gut microbiome diversity, gastrointestinal health, and blood biomarkers. The study will involve 12 participants consuming the test product five times per week, with questionnaires, microbiome testing, blood testing, and waist measurements collected at defined timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female
* Be aged 21-44.
* Anyone currently experiencing issues regarding all of the following:
* Struggling to balance taste with health and convenience.
* Struggling to eat healthy due to a busy lifestyle.
* Self-reported poor gut health (including bloating, abdominal discomfort, and gas).
* Anyone who is generally healthy - does not live with any uncontrolled chronic disease.
* If taking oral over-the-counter supplements or herbal remedies targeted at gut health, blood sugar, and overall health and well-being, has been consistently taking these for at least 3 months prior to starting the study, and is willing to maintain this routine for the study duration.
* Not planning on introducing any products or any new forms of prescription medication or supplements that target gut health, blood sugar, or overall health and well-being for the study duration.
* Anyone willing to maintain their current diet, sleep pattern, and activity levels for the duration of the trial.
* Anyone who has tried pasta alternatives in the past (e.g., made of chickpeas, lentils, beans, etc.) or, if not, is open to trying them.
* Anyone with access to a 3-quart pasta pot that can be used 5 times weekly.
* Resides in the United States.
* Not currently partaking in another research study and will not be partaking in any other research study for the next 12 weeks and at any point during this study's duration.

Exclusion Criteria:

* Has been diagnosed with Type 1 or Type 2 diabetes.
* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone with known severe allergic reactions.
* Anyone with any allergies or sensitivities to any of the study product ingredients.
* Any women who are pregnant, breastfeeding, or trying to conceive (or who will be at any point during the study period).
* Anyone unwilling to follow the study protocol.
* Anyone who has undergone any surgeries or invasive treatments in the last six months.
* Anyone planning to undergo any surgeries or invasive treatments during the study period.
* Anyone with a known history of severe digestive disorders like acid reflux, irritable bowel syndrome (IBS), irritable bowel disease (IBD), Crohn's disease, or gastrointestinal tract surgeries.
* Anyone with a history of substance abuse.
* Anyone who eats a pasta alternative (like chickpea pasta) one or more times per week.
* Follows a specific diet, such as ketogenic, paleo, or gluten-free

Ages: 21 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiome diversity | Baseline and Week 12
  Gut microbiome diversity will be assessed using microbiome testing of stool samples. This outcome will evaluate the effect of the intervention on microbial community richness and composition.
Change in gastrointestinal symptoms using the Gastrointestinal Symptom Rating Scale (GSRS) | Baseline, Week 4, Week 8, and Week 12
  Assessed using the GSRS to evaluate symptoms such as bloating and abdominal discomfort.
Change in blood biomarkers regarding Hemoglobin A1C | Baseline and Week 12
  Measured via blood tests including Hemoglobin A1C with eAG.
Change in blood biomarkers regarding CMP-14 | Baseline and Week 12
  Measured via blood tests including CMP-14, lipid panel, and serum iron to assess metabolic and cardiovascular health indicators.
Change in stool quality using the Bristol Stool Scale (BSS) | Baseline, Week 4, Week 8, and Week 12
  Assessed using the BSS to evaluate stool consistency and form.

SECONDARY OUTCOMES:
Participant-reported perceptions of gut and overall health | Baseline, Week 4, Week 8, and Week 12
  Evaluated through self-reported questionnaires on perceived gut health, weight management, bloating, confidence in clothes, and overall well-being.
Change in waist circumference | Baseline, Week 4, Week 8, and Week 12
  Participants will self-measure and report waist circumference to assess changes in central adiposity over the course of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States